CLINICAL TRIAL: NCT01263184
Title: Längsschnittstudie Zur Belastungsinduzierten Anpassung, Schädigung Oder Degeneration Der Schulter Bei Rollstuhlathleten/-Innen
Brief Title: Symptoms of Degeneration in Shoulder of Wheelchair-users
Acronym: Sodisow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Prof. Dr. Uwe Tegtbur, Institute of Sportsmedicine
Other Study IDs: 5442 - Az 070402/0911
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-11

CONDITIONS: Degeneration; Shoulder Pain
Keywords: shoulder; strength; quality of life
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- sportive wheelchair users
- sportive non disabled
- non sportive wheelchair users

SUMMARY:
The studies object is to evaluate the degeneration of overhead sports in wheelchair-using athletes. It is assumed that wheelchair users do have more symptomatic shoulder pain compared to non disabled athletes.

DETAILED DESCRIPTION:
The force on the shoulder joint is high in handicapped people that are using wheelchairs. The prevalence of chronic shoulder pain for wheelchair-users is as high as 50-80%. Especially paraplegia developed in adult years is predisposed for shoulder pain. The reason is in the short adaption time of the tissue. Dysbalance musculature at the shoulder joint conveys chronic pain. The risk of chronic shoulder pain is rising for wheelchair-users, caused by the lack of recovery-time. After exercising wheelchair users depend on their shoulders in order to manage their daily living. The request of this study is to identify the determinants of shoulder pathologies. Precocious findings in pathologic changes of MRI scans, muscular dysbalance, clinical tests and/or ultrasound-scans lead to certain conclusions. The results should be used to get long-term disorder free situations for sportive wheelchair users.

Scientific background: International publications show relatively uniform results. Paraplegic people and non disabled high performance athletes in overhead sports show cumulative pathologic findings in MRI scans. There is only a minor correlation between MRI findings and clinical symptoms. It is not known how heavy the impact of MRI findings to develop a long term disorder of the shoulder of wheelchair users is. Isokinetic power measurement is a adequate examination of paraplegic people to evaluate the function of the shoulder.

Findings in non disabled high performance athletes: 40% of the asymptomatic high performance athletes in overhead sports show pathologies of their rotator cuff in the dominant arm in MRI (0% in the non dominant arm) (Connor et al. 2003). 10 asymptomatic College Baseball player went through clinical and MRI examination (Halbrecht et al. 1999). It showed pathologic findings the rotator cuff of the dominant side in 7 out of 10 cases. The findings in MRI correlated neither to symptoms nor to the level of instability.

30 asymptomatic athletes out of 52 long distance kayakers were examined with shoulder MRI (Hagemann et al. 2004). 13 asymptomatic kayaker showed pathologic findings in MRI. The authors concluded, that objective MRI findings and subjective discomfort is not highly correlated.

30 high performance handball players showed low correlation between MRI findings and clinical symptoms (Jost et al. 2005). 93% did have pathologic MRI findings, but only 37% were symptomatic.

These studies eliminate, that the clinical symptoms and the subjective impressions, which come up in the career of athletes are not well diagnosed by MRI. Statements about long term effects of rotator cuff tears can not be made. Kelly et al. provided evidence of rotator cuff tears in MRI of 12 non sportive people. 6 of them were symptomatic, 6 were not symptomatic. The subjects that were symptomatic showed lower activation of M. suprascapularis and higher activation of M. trapezius, M. supraspinatus and infraspinatus in EMG diagnosis. In spite of comparable MRI results asymptomatic subjects showed different patterns of innervation of the rotator cuff, than symptomatic subjects. This could lead to a development of muscular dysbalance or longterm defects in the asymptomatic patient. 14 Baseball players, who had no shoulder injury at their shoulder, got MRI scans (Miniaci et al. 2002). 22 of the 28 examined shoulders showed pathologic findings at the labrum. 10 of these athletes were asymptomatic. This is another example of the considerable difference in the felt discomfort and the MRI findings. This statement is not focusing on long term disorders.

MRI examinations in paraplegics: Escobedo et al. did a study in which they examined 26 symptomatic paraplegics with MRI scans on their shoulders. The MRI findings were compared with 17 non disabled subjects, who had symptomatic shoulders as well (Escobedo et al. 1997). 73% of the symptomatic paraplegics (59% of the non disabled) showed rotator cuff tears or following disorders in the MRI scan. 38% of the injured were multiple disorders.

Boninger et al. compared the force input on the wheelchair with MRI findings in 14 paraplegics, who were in average 33 years old. The subjects were asymptomatic and without previous shoulder injuries (Boninger et al. 2003). In intervals of 2 years MRI scans were made. The subjects participated in the study in average 10 years after injury of the spine.

ELIGIBILITY:
Inclusion Criteria:

* capability of doing sports

Exclusion Criteria:

* incapability of doing sports

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: wheelchair users, sportiv people
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-11

PRIMARY OUTCOMES:
Maximum strength measured in isokinetic power measurement | 2 hours

SECONDARY OUTCOMES:
questionnaire: wheelchair users pain index and constant score | 15 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sportsmedicine, Hanover, Lower Saxony, Germany